CLINICAL TRIAL: NCT06057116
Title: The Effect of Massage and Acupressure on Labor Pain and Birth Satisfaction
Brief Title: The Effect of Massage and Acupressure on Labor Pain
Acronym: Neu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Çağla Taş, Chief Investigator Midwife Çağla Taş, Near East University, Turkey
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: YDU/2022/105-1587; YDU/2022/105-1587 (Other Grant/Funding Number: Near East University)
Record Dates: First submitted 2023-08-26; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Labor Pain
Keywords: Massage; acupressure; labor pain; birth satisfaction
MeSH Terms: conditions — Labor Pain | interventions — Massage; Acupressure

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- massage (Experimental): Massage was applied to people who were hospitalized in the obstetrics ward of the pregnant woman, had a single fetus, awaiting spontaneous delivery, had no pregnancy complications, had no systemic disease, and agreed to voluntarily participate in the study.
  Interventions: Other: massage
- acupressure (Experimental): Acupressure for pregnant women who are hospitalized in the obstetrics service, have a single fetus, expect spontaneous delivery, do not have pregnancy complications, do not have any systemic disease, and agree to voluntarily participate in the study.
  Interventions: Other: massage
- control group (No Intervention): No intervention was performed on the patients who were hospitalized in the obstetrics service of the pregnant woman, had a single fetus, awaiting spontaneous delivery, had no pregnancy complications, had no systemic disease, and agreed to voluntarily participate in the study.

INTERVENTIONS:
Other: massage — Massage and acupressure were applied when cervical dilatation was 3-4, 5-7 and 8-10 cm in latent active and transitional phases.
  Other Names: Acupressure
  Arms: acupressure; massage

SUMMARY:
This research was conducted in accordance with the experimental research design to determine the effect of acupuncture and massage, which are non-pharmacological methods used in the treatment of labor pain, on the latent, active and transition stages of the first stage of labor. On labor pain and birth satisfaction. Burhan Nalbantoğlu State Hospital and Near East Hospital. There are three groups in the research sample: acupuncture, massage and control groups. A total of 66 people were reached, 22 people in each group. Massage and acupuncture were applied to the intervention groups, while pregnant women in the control group were not intervened other than routine hospital practices. Cervical dilatation was applied for 3-4, 5-7 and 8-10 cm, and massage was applied for 10 minutes each, for a total of 30 minutes. When cervical dilatation was 3-4, 5-7 and 8-10 cm, acupressure was applied for 1 minute each. The pain level perceived by the pregnant woman was evaluated with the Visual Comparison Scale (VAS), and her satisfaction with the birth was evaluated with the Birth Satisfaction Scale (DME). In comparing the Birth Satisfaction Scale scores and Postpartum Pain VAS Scores, the normal distribution of the data was examined with the Kolmogorov-Smirnov test, Shapiro-Wilk test and skewness-kurtosis values and it was determined that it showed a normal distribution, ANOVA was applied. Tukey test was used in further analysis for comparisons. ANCOVA was applied to compare the amount of pain changes at the beginning and end of the latent, active and transition phases according to participant groups.

DETAILED DESCRIPTION:
The research will be carried out at the Near East Hospital and Nicosia Burhan Nalbantoğlu State Hospital, Gynecology Service. The research will be carried out experimentally, 2 experiments (massage group and acupressure group) and 1 control group will be formed. 95% confidence for the study to be performed with statistically 90% power It was calculated that 22 pregnant women should be given acupressure, 22 pregnant women should be given acupressure and 22 pregnant women should be in the control group with a 5% margin of error. sample size G*Power (Version 3.1.9.2 for Mac) software was used for calculation. Of the pregnant women to be included in the experimental groups; It is planned to be performed with women over the age of 18 and under the age of 35 who are hospitalized in the Gynecology Service of the Near East University Hospital, are at term, have a single fetus, are expected to have spontaneous delivery, do not have pregnancy complications or systemic diseases, and agree to participate in the study. With the volunteer participants who meet these conditions, the study will continue until the number of births is completed. In order to reduce the pain experienced during labor, acupressure will be applied in the first stage of labor, at the end of the latent, active and transitional phases, cervical dilation will be applied for 30 minutes at 3-4, 5-7, 8-10 cm intervals.

In the study, the Visual Analog Scale (VAS) will be used in the evaluation of labor pain. VAS; It is helpful in the broad definition of labor pain. VAS is a horizontally or vertically drawn It is a 10 cm long ruler that says no pain at one end and excruciating pain at the other end. It is thought to be the most appropriate scale among one-dimensional scales in determining the severity of pain, since it gives quick results, is easy and understandable, and is not guided by numbers. Visual Analog Scale is extremely simple, efficient, It is a pain intensity measurement method that can be repeated and requires minimal tools. The Birth Satisfaction Scale (DME) will be used to assess birth satisfaction. DME is a Likert-type scale consisting of 30 questions. The score that can be obtained from the scale varies between 30-150 points. As the score obtained from the scale increases, the satisfaction with the birth increases. VAS scores will be evaluated a total of 3 times at all these stages to assess pain. In the same way, the massage will be evaluated with the VAS score by applying it for 30 minutes in 3 phases. Finally, by making sure that the woman is resting in the postpartum period, a 30-item questionnaire was used to measure her satisfaction with her birth experience.

"Birth Satisfaction Scale" will be filled. The original "Birth Satisfaction Scale (BSS)" was developed in 2009 by Caroline Hollins. Turkish validity and reliability study was conducted by Coşar Çetin F. et al. in 2015. Responses to this 5-point Likert-type scale; Strongly Agree 5; Agree 4; I'm undecided 3; disagree 2; Strongly Disagree Scoring as 1. In scale items; 4, 8, 12, 15, 16, 17, 19, 20, 21, 23, 25 and 29 are scored as reverse items. The total number of points to be taken from the scale varies between 30 and 150 points. The sub-themes in the scale were quality of care, birth environment, adequate support.

ELIGIBILITY:
İnclusion: Having a single fetus, Expecting spontaneous birth, Without Pregnancy Composition, No systemic disease, Those who voluntarily agreed to participate in the research.

Exclusion: With systemic disease multiple pregnancies People who do not want to participate in the research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Skala-VAS | 1 year
  The VAS is a 10 cm long ruler drawn horizontally or vertically with the words "no pain" at one end and "unbearable pain" at the other end.

SECONDARY OUTCOMES:
Birth Satisfaction Scale | 1 year
  The Birth Satisfaction Scale is a Likert-type scale consisting of 30 questions. The score that can be obtained from the scale varies between 30-150 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Çağla Taş, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No